CLINICAL TRIAL: NCT02576860
Title: A Phase 3, Randomized, Vehicle-Controlled, Double-Blind, Multicenter Study to Evaluate the Safety and Efficacy of Once-Daily CLS001 Topical Gel Versus Vehicle Administered for 12 Weeks to Subjects With Papulopustular Rosacea With a 4 Week Follow-up Period
Brief Title: Study to Evaluate the Safety and Efficacy of a Once-Daily CLS001 Topical Gel Versus Vehicle
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-005
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Results first posted 2022-07-08 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Omiganan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): CLS001 (Omignan) gel applied once daily
  Interventions: Drug: CLS001 (Omiganan)
- Vehicle Gel (Placebo Comparator): Vehicle gel applied once daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CLS001 (Omiganan) — Topical gel
  Arms: Treatment
Drug: Vehicle — Vehicle gel
  Arms: Vehicle Gel

SUMMARY:
This study evaluates the safety and efficacy of once-daily application of CLS001 topical gel compared to vehicle gel in subjects with severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male and non-pregnant female subjects, 18 years of age or older.
2. A diagnosis of papulopustular rosacea with ≥30 inflammatory facial lesions at Baseline. Subjects must have no more than 2 nodular lesions, at Baseline.
3. Subjects with the presence of telangiectasia at Baseline.
4. Subjects with an erythema score of at least 2 on the Investigator Assessment of Erythema scale at Baseline.
5. Subjects with severe rosacea on the Investigators Global Assessment scale at Baseline.

Exclusion Criteria:

1. Subjects with steroid rosacea or subtype 3 (phymatous rosacea).
2. Subjects with nodular rosacea.
3. Standard exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02-27 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (20):
  - Fort Smith, Arkansas
  - Rogers, Arkansas
  - Manhattan Beach, California
  - Oceanside, California
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Miami, Florida
  - Plainfield, Indiana
  - Watertown, Massachusetts
  - Omaha, Nebraska
  - Verona, New Jersey
  - New York, New York
  - Stony Brook, New York
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fort Washington, Pennsylvania
  - Charleston, South Carolina
  - Arlington, Texas
  - San Antonio, Texas
- Australia (4):
  - Phillip, Australian Capital Territory
  - Kogarah, New South Wales
  - Liverpool, New South Wales
  - Box Hill, Victoria
- Canada (4):
  - Surrey, British Columbia
  - Courtice, Ontario
  - Peterborough, Ontario
  - Windsor, Ontario
- France (3):
  - Grenoble
  - Nantes
  - Quimper
- Germany (10):
  - Berlin
  - Bochum
  - Bonn
  - Cologne
  - Friedrichshafen
  - Hamburg
  - Lingen
  - Mönchengladbach
  - Osnabrück
  - Schweinfurt
- Nijmegen, Netherlands
- Auckland, New Zealand
- Halmstad, Sweden
- United Kingdom (3):
  - Bradford, England
  - Birmingham
  - London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 sites in the USA, Canada, Australia/New Zealand, and durope from December 2015 to February 2017.
Period: Overall Study
Arm/Group | Treatment | Vehicle Gel
Started | 136 | 127
Completed | 111 | 103
Not Completed | 25 | 24
Not completed — Adverse Event | 6 | 6
Not completed — Lost to Follow-up | 5 | 7
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 13 | 8
Not completed — Disallowed medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Vehicle Gel | Total
Number analyzed (Participants) | 136 | 127 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 109 | 100 | 209
  >=65 years | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (14.06) | 52.4 (13.66) | 51.8 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 70 | 155
  Male | 51 | 57 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 35
  Not Hispanic or Latino | 118 | 110 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 130 | 122 | 252
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 64 | 129
Total Inflammatory Lesion Count [Mean (Standard Deviation); unit: lesion count] — Defined as the total number of papules and pustules.
  lesion count | 53.1 (24.78) | 51.0 (19.42) | 52.1 (22.34)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Absolute Change in Inflammatory Lesion Count
Description: Absolute change in inflammatory lesion count from baseline to Week 12.
Time Frame: 12 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Lesions | -19.8 (2.29) | -20.9 (2.36)
Statistical Analysis 1: Comparison: Treatment vs Vehicle Gel; Test type: Superiority; p = 0.799, ANCOVA

2. Primary Outcome: Efficacy IGA: 2 Grade Reduction
Description: Proportion of Subjects Who Achieved 2 Grade IGA Reduction at Week 12. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 12 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Percentage of Subjects | 24.6 | 25.6
Statistical Analysis 1: Comparison: Treatment vs Vehicle Gel; Test type: Superiority; p = 0.858, Cochran-Mantel-Haenszel

3. Secondary Outcome: Efficacy The Absolute Change in Inflammatory Lesions
Description: The absolute change in inflammatory lesions from baseline to Week 9.
Time Frame: 9 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Lesions | -21.6 (2.23) | -20.9 (2.3)

4. Secondary Outcome: Efficacy The Absolute Change in Inflammatory Lesions
Description: The absolute change in inflammatory lesions from baseline to Week 6.
Time Frame: 6 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: Lesions
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Lesions | -16.2 (1.96) | -19.8 (2.06)

5. Secondary Outcome: Efficacy IGA: 2 Point Reduction
Description: Proportion of Subjects Who Achieved 2 Grade IGA Reduction at Week 9. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 9 Weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Percentage of Subjects | 23.7 | 21.6

6. Secondary Outcome: Efficacy IGA: 2 Point Reduction
Description: Proportion of Subjects Who Achieved 2 Grade IGA Reduction at Week 6. IGA scores are from 0 to 5 (Clear, Almost Clear, Mild, Moderate and Severe).
Time Frame: 6 Weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Treatment | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Percentage of Subjects | 15.2 | 15.9

7. Other Pre Specified Outcome: Safety Adverse Events
Description: Subjects with 1 or more treatment-related Treatment-Emergent Adverse Events
Time Frame: 12 weeks
Population: The 'Intent-to-treat' (ITT) analysis population included all randomized subjects.
Measure: Count of Participants; unit: Participants
Groups:
- CLS001 (Omignan) Gel: CLS001 (Omignan) gel applied once daily
  CLS001 (Omiganan): Topical gel
Arm/Group | CLS001 (Omignan) Gel | Vehicle Gel
Number analyzed (Participants) | 136 | 127
Participants | 19 | 17

ADVERSE EVENTS:
Time Frame: 115 Days
Arm/Group | Treatment | Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/127
Serious Adverse Events (participants affected / at risk) | 1/136 | 0/127
Other Adverse Events (participants affected / at risk) | 47/136 | 36/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=136) | Vehicle Gel (N=127)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=136) | Vehicle Gel (N=127)
Viral upper respiratory tract infection (Infections and infestations) | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Bronchitis (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 0 | 4
Application site pain (General disorders) | 9 | 2
Application site erythema (General disorders) | 4 | 5
Application site pruritus (General disorders) | 3 | 5
Headache (Nervous system disorders) | 9 | 6
Rosacea (Skin and subcutaneous tissue disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT02576860/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT02576860/SAP_001.pdf